CLINICAL TRIAL: NCT02452619
Title: Brain Angiogenesis Induced by Hyperbaric Oxygen Therapy Can be Visualized by Perfusion MRI in Brain Injury Patients
Brief Title: MRI Brain Changes Induced by Hyperbaric Oxygen Therapy in Brain Injury Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Dr Sigal Tal, Assaf-Harofeh Medical Center
Other Study IDs: 0030-15-ASF
Record Dates: First submitted 2015-04-15; First posted 2015-05-22 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Hyperbaric Oxygen Therapy; Mild Cognitive Impairment
Keywords: Hyperbaric oxygen therapy; brain trauma; cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction; Brain Injuries, Traumatic | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Brain trauma: Patients with chronic brain injury that have been treated with Hyperbaric oxygen therapy and underwent MRI imaging and cognitive tests before and after the treatment
  Interventions: Other: Hyperbaric oxygen therapy

INTERVENTIONS:
Other: Hyperbaric oxygen therapy — Hyperbaric oxygen therapy

SUMMARY:
In our institute there is ongoing treatment of brain injury patients with Hyperbaric oxygen therapy. These patients undergo neuro-cognitive function tests in addition to brain imaging studies before and after treatment.

The aim of this study was to evaluate the perfusion and microstructure changes seen in MRI in addition to the cognitive tests before and after the treatment.

DETAILED DESCRIPTION:
Retrospective analysis of patients suffering from chronic neuro-cognitive damage due to TBI treated at Sagol center for hyperbaric medicine and research, Assaf Harofeh Medical Center, Israel

Patients included if they had at least two perfusion MRIs + DTI and two neurocognitive tests, before and after Hyperbaric Oxygen Therapy (HBOT). The study was approved by the institutional review board of the hospital.

Patients are treated with 50-70 daily hyperbaric sessions, 5 days per week. Each session consists of 60 minutes exposure to 100% oxygen at 1.5 ATA.

All patients that underwent MRI before and after HBOT. The MRI protocol included DSC, DCE, DTI, FLAIR, T2 and SWI.

MRI scans sequences parameters:

* DSC: 50 T2*-weighted gradient-echo echo planar imaging (EPI) volumes were acquired, 2 repetitions before a bolus injection of Gadolinium-DTPA (Gd-DTPA), 48 repetitions after injection of Gd-DTPA. Sequence parameters: TR=2,300 ms, TE= 40ms, flip angle = 30°, voxel size = 1.8 x1.8, Matrix = 128x128, No. of slices = 25, Slice thickness = 3.9 mm.

* DCE: three T1 weighted Fast Low Angle SHot (FLASH) volumes were acquired with different flip angles (2, 7 and 15 degrees) followed by 70 dynamic T1 weighted FLASH volumes with flip angle of 15 degrees after bolus injection of Gd-DTPA. Sequence parameters: before injection: TR=4.09, after injection - TR=4.86 ms, TE= 1.76 ms, Voxel size = 1.5x1.5, Matrix = 192X192, No. of slices = 26, Slice thickness = 3.5mm.
* DTI: 30 diffusion weighted images were scanned with different gradient directions (b=1000) and one volume without diffusion weighting, with the following parameters: TR=10,300 ms, TE=89 ms, Voxel size = 1.8X1.8, Matrix = 128 X 128, No. of slices = 63, Slice thickness = 2.2mm

ELIGIBILITY:
Inclusion Criteria:

* Patients included if they had at least two perfusion MRIs + DTI and two neurocognitive tests, before and after Hyperbaric Oxygen Therapy (HBOT).

Exclusion Criteria:

* did no complete treatment or did not complete examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective analysis of patients suffering from chronic neuro-cognitive damage treated at Sagol center for hyperbaric medicine and research, Assaf Harofeh Medical Center, Israel from September 2013 .
  Patients included if they had at least two perfusion MRIs + DTI and two neurocognitive tests, before and after Hyperbaric Oxygen Therapy (HBOT). Treatment was approved by the institutional review board of the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Perfusion MRI changes | Before and after treatment. Treatment is approximately 3 months.
Microstructure changes (DTI) | Before and after treatment. Treatment is approximately 3 months.

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Assaf-Harofeh Medical Center, Ẕerifin, Israel
  - Assaf-Harofeh Medical Center, Ẕerifin